CLINICAL TRIAL: NCT02229149
Title: Randomized Phase II Trial of Chemotherapy of Physician's Choice Plus Trastuzumab Versus Chemotherapy of Physician's Choice Plus Trastuzumab Plus Pertuzumab In Women With Pretreated, HER2-Overexpressing Metastatic Breast Cancer (MBC)
Brief Title: Phase 2 Study of Standard Chemotherapy With Trastuzumab, Plus or Minus Pertuzumab, for Pre-treated Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: per Sponsor request
Sponsor: US Oncology Research (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13011; ML29212 (Other: Genentech, Inc.)
Record Dates: First submitted 2014-08-27; First posted 2014-08-29 (Estimated); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Breast Neoplasms; Malignant Tumor of the Breast
Keywords: breast cancer; metastatic breast cancer; HER2+ breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; pertuzumab; Vinorelbine; Paclitaxel; 130-nm albumin-bound paclitaxel; Docetaxel; Capecitabine; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Triple Therapy (Experimental): Physician's choice of chemotherapy plus trastuzumab plus pertuzumab
  * trastuzumab, given as a loading dose of 8 mg/kg intravenously (IV, or through the vein) on Day 1 followed by 6 mg/kg IV every 3 weeks thereafter, AND
  * physician's choice of chemotherapy:
    1. Vinorelbine 25 mg/m2 IV weekly times 3 with 1 week off; OR
    2. Paclitaxel 80 mg/m2 IV weekly times 3 with 1 week off; OR
    3. Nab-Paclitaxel 100 mg/m2 IV weekly times 3 with 1 week off; OR
    4. Docetaxel 75 mg/m2 IV every 3 weeks; OR
    5. Capecitabine 1500 mg by mouth twice a day (PO BID) 14 days on and then 7 days off.
  * AND pertuzumab given as a loading dose of 840 mg IV on Day 1 followed by 420 mg IV every 3 weeks.
  Interventions: Drug: Trastuzumab; Drug: Pertuzumab; Drug: Vinorelbine, Paclitaxel, Nab-Paclitaxel , Docetaxel, Capecitabine
- Double Therapy (Active Comparator): Physician's choice of chemotherapy plus trastuzumab
  * trastuzumab, given as a loading dose of 8 mg/kg intravenously (IV, or through the vein) on Day 1 followed by 6 mg/kg IV every 3 weeks thereafter, AND
  * physician's choice of chemotherapy:
    1. Vinorelbine 25 mg/m2 IV weekly times 3 with 1 week off; OR
    2. Paclitaxel 80 mg/m2 IV weekly times 3 with 1 week off; OR
    3. Nab-Paclitaxel 100 mg/m2 IV weekly times 3 with 1 week off; OR
    4. Docetaxel 75 mg/m2 IV every 3 weeks; OR
    5. Capecitabine 1500 mg PO BID 14 days on and then 7 days off.
  Interventions: Drug: Trastuzumab; Drug: Vinorelbine, Paclitaxel, Nab-Paclitaxel , Docetaxel, Capecitabine

INTERVENTIONS:
Drug: Trastuzumab — Treatment for all patients will consist of trastuzumab, given as a loading dose of 8 mg/kg IV on Day 1 followed by 6 mg/kg IV every 3 weeks thereafter.
  Patients randomized to the chemotherapy plus trastuzumab arm (without pertuzumab) can receive trastuzumab 6 mg/kg IV every 3 weeks if they are receiving docetaxel or capecitabine on a 3-week cycle, or 4 mg/kg IV every 2 weeks if they are receiving vinorelbine, paclitaxel, or nab-paclitaxel on a 4-week cycle. The loading dose for all patients remains 8 mg/kg.
  For patients randomized to the chemotherapy plus trastuzumab plus pertuzumab arm, both trastuzumab and pertuzumab need to be administered every 3 weeks regardless of which chemotherapy agent they are receiving.
  Other Names: Herclon, Herceptin
Drug: Pertuzumab — pertuzumab given as a loading dose of 840 mg IV on Day 1 followed by 420 mg IV every 3 weeks.
  Other Names: 2C4; Perjeta; Omnitarg
  Arms: Triple Therapy
Drug: Vinorelbine, Paclitaxel, Nab-Paclitaxel , Docetaxel, Capecitabine — physician's choice of chemotherapy:
  * Vinorelbine 25 mg/m2 IV weekly times 3 with 1 week off; OR
  * Paclitaxel 80 mg/m2 IV weekly times 3 with 1 week off; OR
  * Nab-Paclitaxel 100 mg/m2 IV weekly times 3 with 1 week off; OR
  * Docetaxel 75 mg/m2 IV every 3 weeks; OR
  * Capecitabine 1500 mg by mouth twice a day (PO BID) 14 days on and then 7 days off.
  Other Names: Navelbine; Abraxane; Taxol; Taxotere; Docecad; Xeloda

SUMMARY:
This randomized phase 2 study will seek to determine the effectiveness of chemotherapy (physician's choice of vinorelbine, taxane [paclitaxel, docetaxel or nab paclitaxel] or capecitabine) plus trastuzumab vs chemotherapy (physician's choice) plus trastuzumab plus pertuzumab in women with HER2-overexpressing metastatic breast (MBC) that has been previously treated with ado-trastuzumab emtansine (T-DM1) in the metastatic setting.

DETAILED DESCRIPTION:
The current preferred first-line therapy for patients with HER2-overexpressing metastatic breast cancer (MBC) is a taxane plus trastuzumab plus pertuzumab, based on results from the CLEOPATRA trial. For patients with disease that has progressed on trastuzumab and a taxane, ado-trastuzumab emtansine (T-DM1) was recently approved based on results from the EMILIA trial showing superiority in this setting compared with capecitabine plus lapatinib. However, the standard for first-line therapy may change again in the near future, when results become available from the MARIANNE trial, which is evaluating T-DM1 alone or in combination with pertuzumab as upfront therapy. Two important questions that may be raised by the findings of this study are whether pertuzumab is effective as second- or later-line therapy following single-agent T-DM1, and whether pertuzumab administered beyond progression on prior pertuzumab therapy is of clinical benefit as trastuzumab has been proven to be.

The study will seek to determine the efficacy of chemotherapy (physician's choice of vinorelbine, taxane [paclitaxel, docetaxel or nab paclitaxel] or capecitabine) plus trastuzumab vs chemotherapy (physician's choice) plus trastuzumab plus pertuzumab in women with HER2-overexpressing MBC that has been previously treated with T-DM1 in the metastatic setting.

We hypothesize that the addition of pertuzumab to trastuzumab plus chemotherapy will improve median progression-free survival (PFS), compared to trastuzumab plus chemotherapy alone, as second- or later-line therapy in patients who have received prior T-DM1. Patients will be stratified according to whether they have received prior pertuzumab versus not. We will also explore whether continuing treatment with pertuzumab in patients who have been previously treated with pertuzumab improves PFS.

ELIGIBILITY:
Inclusion Criteria:

1. Female, Age ≥ 18 years
2. Histologic or cytologic confirmation of human epidermal growth factor receptor 2 (HER2)-positive breast cancer according to most recent biopsy (local testing permitted)
3. Measurable or evaluable metastatic disease by Response Evaluation Criteria in Solid Tumors (RECIST) (v1.1)
4. Previous treatment with ado-trastuzumab emtansine (T-DM1) for metastatic disease

   a. Prior therapy with pertuzumab is allowed but not required
5. At least 1 but no more than 3 prior chemotherapy regimens for metastatic breast cancer (MBC)
6. Life expectancy > 6 months
7. Eastern Cooperative Group (ECOG) performance status ≤ 2
8. Left Ventricular Ejection Fraction (LVEF) ≥ 50% at baseline as determined by either echocardiogram (ECHO) or Multi Gated Acquisition Scan (MUGA) and within normal limits per institutional guidelines
9. Adequate bone marrow function as indicated by the following:

   1. Absolute Neutrophil Count (ANC) ≥1500/uL (or 1500 per microliter)
   2. Platelets ≥100,000/uL
   3. Hemoglobin >9 g/dL
10. Adequate renal function, as indicated by creatinine <1.5 times upper limit of normal (ULN)
11. Adequate liver function, as indicated by bilirubin <1.5 times ULN
12. Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) <2 x ULN unless liver metastases are present in which case AST and ALT up to 5.x ULN are allowed
13. Negative serum pregnancy test within 72 hours before starting study medications for women of childbearing potential
14. Women of childbearing potential must be willing to use an acceptable form of birth control (ie, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study Note: Women are considered postmenopausal and not of childbearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms), or if they have undergone surgical sterilization.
15. Signed informed consent obtained prior to any screening procedures.

Exclusion Criteria:

Patients will be excluded from the study based on the following criteria:

1. Prior treatment in the metastatic setting with the agent chosen as physician's choice of chemotherapy
2. Active infection
3. Uncontrolled central nervous system metastases, defined as clinical or radiologic evidence of progression of brain metastases or clinical signs of leptomeningeal disease

   a. Patients with treated brain metastases are eligible provided they do not have clinical or radiologic evidence of disease progression and have been off of dexamethasone for at least 3 weeks
4. Patient is pregnant or lactating
5. Prior chemotherapy within the last 3 weeks (last 6 weeks for nitrosureas/mitomycin)
6. Prior radiation therapy within the last 2 weeks; prior radiation therapy to indicator lesion (unless objective disease recurrence or progression within the radiation portal has been documented since completion of radiation).
7. Requirement for chronic steroid therapy with a requirement for > 5mg/day of prednisone or the equivalent.

   a. Treatment with physiologic doses of hydrocortisone up to 20 mg daily (QD) is allowed.
8. Requirement for immunosuppressive therapy, such as those used to treat autoimmune disease.
9. Concomitant malignancies or previous malignancies within the last 3 years, with the exception of adequately treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.
10. History of significant cardiac disease, cardiac risk factors or uncontrolled arrhythmias
11. Ejection fraction <50% or below the lower limit of the institutional normal range, whichever is lower
12. Known hypersensitivity to trastuzumab or pertuzumab
13. Serious medical or psychiatric limitations likely to interfere with participation in this study.
14. Symptomatic intrinsic lung disease or extensive tumor involvement of the lungs, resulting in dyspnea at rest or requiring supplemental oxygen
15. Patient is currently part of or has participated in any clinical trial of an investigational agent within 1 month prior to enrollment in this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2022-01 (Actual); Study Completion 2022-01 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 2 years
  The primary objective of this study is to compare progression-free survival (PFS [also known as time to disease progression]) with the addition of pertuzumab to trastuzumab plus physician's choice of chemotherapy versus trastuzumab plus physician's choice of chemotherapy in patients who have previously received treatment with ado-trastuzumab emtansine (TDM1) for HER2+ metastatic breast cancer.

SECONDARY OUTCOMES:
Progression-free survival (PFS) in patients (pts) with prior pertuzumab | 2 years
  To assess PFS with the addition of pertuzumab to trastuzumab plus physician's choice of chemotherapy in patients who have received prior pertuzumab;
Progression-free survival (PFS) in pts with prior chemotherapy | 2 years
  To compare median PFS with the addition of pertuzumab to trastuzumab plus physician's choice of chemotherapy in patients who have received 1 vs 2-3 prior chemotherapy regimens for metastatic disease;
Number of patients with complete and partial responses | 2 years
  To compare the objective response rates (ORR; complete response [CR] plus partial response [PR]) between the two treatment arms;
Overall survival | 2 years
  To assess overall survival (OS) in each of the treatment arms;
Number of adverse events and serious adverse events | 2 years
  To assess the safety of pertuzumab in combination with trastuzumab and physician's choice of chemotherapy (vinorelbine, paclitaxel, nab-paclitaxel, docetaxel, or capecitabine).

CONTACTS AND LOCATIONS:
Overall Officials: Neelima Denduluri, MD, Principal Investigator — US Oncology Research, McKesson Specialty Health
Locations (1):
- 19 Sites, Multiple Locations, Texas, United States